CLINICAL TRIAL: NCT04272385
Title: Defining Core Outcome Sets in Trigeminal Neuralgia
Acronym: TRINCOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Rosetrees Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 17/0901
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Trigeminal Neuralgia
Keywords: trigeminal neuralgia; treatment outcomes; patient reported outcome measures
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Focus Group: Qualitative research done with a group of patients with TN. Patients will describe their experience of living with the disease and what outcomes of treatment they consider to be important.
  Interventions: Other: Observational
- Delphi survey: Group of relevant stakeholders - patients, clinicians and researchers will rate the outcomes of treatment in a 3 round Delphi survey.
  Interventions: Other: Observational
- Consensus meeting: Group of relevant stakeholders - patients, clinicians and researchers will rate the outcomes of treatment and finalise the COS for Trigeminal Neuralgia.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
The aim of this study is to determine what patients with trigeminal neuralgia (TN), clinicians and researchers in the field, consider to be the most important outcomes to be expected after undergoing treatment for trigeminal neuralgia and how this could be measured in all studies relating to this condition. This would enable different treatments to be compared using the same standards.

DETAILED DESCRIPTION:
Trigeminal Neuralgia (TN) is a rare chronic condition that causes agonizing, unpredictable, short-lasting electric shock-like one-sided facial pain and is commonly provoked by triggers such as light touch. This debilitating chronic pain disorder has a significant impact on the quality of life of patients with increased risk of depression and suicide. The current varied outcome measures make it difficult for patients to make decisions about choice of treatments which was highlighted in a study among 156 United Kingdom (UK) patients with TN who completed an adapted time-trade - off utility measure to ascertain how they valued the potential outcomes from various surgical and medical treatments.

Patients can be managed with a range of anticonvulsants or by several types of neurosurgical interventions. To successfully compare the effectiveness and tolerability of various treatment options data is needed from well designed and conducted randomised controlled trials (RCTs) and prospective cohorts which use the same outcome measures. Apart from pain relief only a handful of other outcome measures have been used. It has to date not been possible to compare medical versus neurosurgical treatments and yet this is one of the most frequently asked patient questions. The impact of complications on ability to return to normal activities and improvement in mental health needs to be determined. The development and implementation of Core Outcome Sets (COS) and measures in clinical practice across the UK and in future trials would allow standardised outcome data, thereby facilitating meta-analysis and thus clinical decision-making.

ELIGIBILITY:
Inclusion Criteria for the focus groups:

* Adult patients (>18ys) diagnosed with trigeminal neuralgia
* Willing to attend a focus group meeting
* Able to give informed consent
* Undergoing management for trigeminal neuralgia

Exclusion Criteria:

* Unable to attend a focus group meeting
* Insufficient English to take part in a group discussion
* Unable to take part in discussions

Inclusion Criteria for the Delphi survey:

* Adult patients (>18ys) diagnosed with trigeminal neuralgia
* Clinicians working in the field of Trigeminal Neuralgia

  * Researchers working in the field of Trigeminal Neuralgia
  * Willing to complete a 3 round Delphi survey
* Able to give informed consent

Inclusion Criteria for the online consensus meeting:

* Adult patients (>18ys) diagnosed with trigeminal neuralgia
* Clinicians working in the field of Trigeminal Neuralgia

  * Researchers working in the field of Trigeminal Neuralgia
  * Able to join an online meeting
  * Have internet access
  * Willing to participate in a discussion with others about the important treatment outcomes in Trigeminal Neuralgia
* Able to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with trigeminal neuralgia and are currently receiving treatment (medical or surgical). Clinicians and researchers working in the field.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Define the trigeminal neuralgia core outcome set | 2020-2022

SECONDARY OUTCOMES:
Identify the instruments to use in the core outcome set | 2020-2022

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Zakrzweska, Professor, Principal Investigator — University College, London
Locations (1):
- The Royal National ENT and Eastman Dental Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.comet-initiative.org/Studies/Details/1123